CLINICAL TRIAL: NCT04465929
Title: Expanded Access - The Safety and Efficacy of Autologous Human Schwann Cell (ahSC) Augmentation of Nerve Autografts After Severe Peripheral Nerve Injury (PNI)
Brief Title: Expanded Access - Autologous Human Schwann Cells in Peripheral Nerve Repair
Status: No longer available | Type: Expanded Access
Sponsor: W. Dalton Dietrich (Other)
Responsible Party: Sponsor-Investigator, W. Dalton Dietrich, Professor, University of Miami
Organization: University of Miami (Other)
Other Study IDs: 20190453-EAP
Record Dates: First submitted 2020-06-25; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Peripheral Nerve Injuries
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Autologous Human Schwann Cells — Schwann cells harvested from the sural nerve and debrided, injured sciatic nerve of the participant will be autologously transplanted along sural nerve autografts wrapped in a collagen matrix

SUMMARY:
Emergency expanded access for a single patient was granted to receive autologous human Schwann cell (ahSC) augmentation of nerve autograft repair after severe peripheral nerve injury (PNI).

ELIGIBILITY:
Inclusion Criteria:

* Persons with severe sciatic nerve injury, brachial plexus injury, and/or major injury at the upper or lower extremity with nerve loss within previous year;
* Peripheral nerve injury with large gap (5 - 10 cm) between healthy nerve endings;

Exclusion Criteria:

* Persons unable to safely undergo an MRI (may include persons with an implanted device or metallic fragments which may interfere with MRI safety);
* Persons with pre-existing conditions that would preclude satisfactory sural nerve harvest (may include amputation or major injury to lower limb, or disease affecting the sural nerve);
* Persons with severe peripheral nerve injury gap length > 10 cm in length;
* Persons with history of radiation or local cancer in area of nerve injury, including primary tumors of the nerve;
* Pregnant women or a positive pregnancy test in those women with reproductive potential prior to transplantation;
* Presence of disease that might interfere with participant

Ages: 16 Years to 16 Years | Sex: Female
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Allan D. Levi, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States